CLINICAL TRIAL: NCT06009809
Title: Blood Velocity Variation in Right Renal and Superior Mesenteric Arteries During Cardio-pulmonary Bypass
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr.ssa Gabriella Arlotta, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4708
Record Dates: First submitted 2022-05-26; First posted 2023-08-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Heart Surgical Procedure
Keywords: cardiopulmonary by-pass; transesophageal echocardiogram; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Surgical Patients: Patients with cardiovascular disease, who must undergo cardiac surgery in extracorporeal circulation with continuous flow
  Interventions: Diagnostic Test: transesophageal echocardiogram

INTERVENTIONS:
Diagnostic Test: transesophageal echocardiogram — To measure mean blood velocity at the level of the right renal and superior mesenteric artery

SUMMARY:
The cardiopulmonary by-pass technique, used in cardiac surgery to obtain a bloodless operating field and an immobile heart, determines important effects on the blood vessel wall, especially when a continuous and non-continuous blood flow is used. In fact, a reduction in Nitric Oxide (NO) production by the endothelium, an increase in systemic vascular resistance and an increased risk of cerebral and renal hypoperfusion have been observed and can result in potential organ damage. Acute kidney injury (AKI) after heart surgery is a major cause of mortality and morbidity. Its incidence varies according to different definitions, but can reach 30%. In some series, 1-5% of patients require renal replacement therapy in the postoperative period presenting a mortality that can reach 50-70%. However, even more limited increases in serum creatinine are associated with worsening prognosis and the risk of chronic kidney disease. The pathophysiology of AKI in cardiac surgery is complex and still partly unknown.Recently a technique has been described that allows to measure the blood velocity in the right renal artery and in the superior mesenteric artery using the transesophageal echocardiogram (TEE); this technique allows to view these arteries and measure the speed of the blood with good precision because the insonation angle (ie the angle formed by the ultrasound flow and the direction of the blood vessel) is adequate. In cardiac surgery, this methodology allows you to monitor blood velocity in the right renal artery and superior mesenteric artery during surgery. Some authors have used it to conduct pilot studies in which the blood velocity values in the renal arteries during cardiac surgery were used to calculate the pulsatility and resistivity indices, as predictors of the risk of postoperative AKI. At present, therefore, despite the fact that TEE is routinely used for monitoring renal perfusion during cardiac surgery, the blood velocity in the renal and mesenteric arteries has been little studied during cardiopulmonary by-pass (CPB) and has never been evaluated during CPB with continuous flow; in particular, the possible variation in blood velocity measured during CPB compared to the baseline values measured before extracorporeal circulation and its correlation with the onset of postoperative renal failure is not known.

DETAILED DESCRIPTION:
The cardiopulmonary by-pass (CPB) technique, used in cardiac surgery to obtain a bloodless operating field and an immobile heart, determines important effects on the blood vessel wall, especially when a continuous and non-continuous blood flow is used. In fact, a reduction in NO production by the endothelium, an increase in systemic vascular resistance and an increased risk of cerebral and renal hypoperfusion have been observed and can result in potential organ damage.

Acute kidney injury (AKI) after heart surgery is a major cause of mortality and morbidity. Its incidence varies according to different definitions, but can reach 30%. In some series, 1-5% of patients require renal replacement therapy (RRT) in the postoperative period presenting a mortality that can reach 50-70%. However, even more limited increases in serum creatinine (sCr) are associated with worsening prognosis and the risk of chronic kidney disease (CKD). The pathophysiology of AKI in cardiac surgery is complex and still partly unknown. It is believed that one of the main causative factors is hypoperfusion and renal hypoxia, in particular of the medullary region; this would result in a vasoconstriction of the afferent arterioles to the glomerulus and a reduction in filtration. Risk factors associated with the increased incidence of AKI include bleeding, use of the aortic pump, excessive cardiopulmonary bypass duration, excessive haemodilution, insufficient pump flow, or insufficient blood pressure. Hypothermia, which also has a protective effect against hypoperfusion and tissue hypoxia, could induce AKI by increasing renal vascular resistance and favoring medullary hypoxia during subsequent rewarming.

In addition to AKI, another complication of cardiac surgery, rarer but associated with a higher mortality, is acute mesenteric ischemia; the most frequent type is non-occlusive mesenteric ischemia (NOMI) which seems to have as a predisposing cause a reduction or maldistribution of splanchnic blood flow and the use of vasoconstrictors.

Recently a technique has been described that allows to measure the blood velocity in the right renal artery and in the superior mesenteric artery using the transesophageal echocardiogram (TEE); this technique allows to view these arteries and measure the speed of the blood with good precision because the insonation angle (ie the angle formed by the ultrasound flow and the direction of the blood vessel) is adequate. In cardiac surgery, this methodology allows you to monitor blood velocity in the right renal artery and superior mesenteric artery during surgery. Some authors have used it to conduct pilot studies in which the blood velocity values in the renal arteries during cardiac surgery were used to calculate the pulsatility and resistivity indices, as predictors of the risk of postoperative AKI. The calculation of these indices, however, requires the use of a pulsatile blood flow to generate a periodic variation of the blood velocity, and they are not evaluable during CPB since the current practice in almost all centers is to use a continuous blood flow. At present, therefore, despite the fact that TEE is routinely used for monitoring renal perfusion during cardiac surgery, the blood velocity in the renal and mesenteric arteries has been little studied during CPB and has never been evaluated during CPB with continuous flow; in particular, the possible variation in blood velocity measured during CPB compared to the baseline values measured before extracorporeal circulation and its correlation with the onset of postoperative renal failure is not known.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* written informed consent
* cardiac surgery with cardiopulmonary bypass (CPB)
* New York Heart Association (NYHA) class I, II, III
* preoperative serum creatinine less than 1.2 mg / dl

Exclusion Criteria:

* contraindications to Trans Esophageal Ultrasound (TEE) based on American Society of Anesthesiologists (ASA) recommendations (esophageal or gastric diseases or previous surgery)
* history of non-coronary arterial pathologies
* atrial fibrillation
* preoperative serum creatinine greater than 1.2 mg / dl • NYHA class IV
* emergency cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients of both sexes, aged> 18 years, with cardiovascular disease, who must undergo cardiac surgery in extracorporeal circulation with continuous flow
Sampling Method: Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of right renal artery mean blood velocities before and during cardiopulmonary by-pass (CPB) | Basal 1: up to 10 minutes after induction of anesthesia and placement of transesophageal probe
  Right renal artery mean blood velocity (cm/sec) before CPB
Comparison of right renal artery mean blood velocities before and during cardiopulmonary by-pass (CPB) | Basal 2: up to 30 minutes after sternotomy in conditions of hemodynamic stability
  Right renal artery mean blood velocity (cm/sec) before CPB
Comparison of right renal artery mean blood velocities before and during cardiopulmonary by-pass (CPB) | CPB 5 min: during CPB, 5 minutes after the end of the first cardioplegia
  Right renal artery mean blood velocity (cm/sec) during CPB
Comparison of right renal artery mean blood velocities before and during cardiopulmonary by-pass (CPB) | CPB 30 min: during CPB, 30 minutes after the end of the first cardioplegia
  Right renal artery mean blood velocity (cm/sec) during CPB
Comparison of right renal artery mean blood velocities before and during cardiopulmonary by-pass (CPB) | CPB 60 min: during CPB, 60 minutes after the end of the first cardioplegia
  Right renal artery mean blood velocity (cm/sec) during CPB

SECONDARY OUTCOMES:
Comparison of superior mesenteric artery mean blood velocities before and during cardiopulmonary by-pass (CPB) | Basal 1: up to 10 minutes after induction of anesthesia and placement of transesophageal probe
  Superior mesenteric artery mean blood velocity (cm/sec) before CPB
Comparison of superior mesenteric artery mean blood velocities before and during cardiopulmonary by-pass (CPB) | Basal 2: up to 30 minutes after sternotomy in conditions of hemodynamic stability
  Superior mesenteric artery mean blood velocity (cm/sec) before CPB
Comparison of superior mesenteric artery mean blood velocities before and during cardiopulmonary by-pass (CPB) | CPB 5 min: during CPB, 5 minutes after the end of the first cardioplegia
  Superior mesenteric artery mean blood velocity (cm/sec) during CPB
Comparison of superior mesenteric artery mean blood velocities before and during cardiopulmonary by-pass (CPB) | CPB 30 min: during CPB, 30 minutes after the end of the first cardioplegia
  Superior mesenteric artery mean blood velocity (cm/sec) during CPB
Comparison of superior mesenteric artery mean blood velocities before and during cardiopulmonary by-pass (CPB) | CPB 60 min: during CPB, 60 minutes after the end of the first cardioplegia
  Superior mesenteric artery mean blood velocity (cm/sec) during CPB
Correlation between mean blood velocity values and hemodynamic parameters: cardiopulmonary by-pass (CPB) blood flow | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between right renal artery mean blood velocity (cm/sec) and CPB blood flow (L/min)
Correlation between mean blood velocity values and CPB blood flow | CPB 30 min: 30 minutes after the end of the first cardioplegia, during CPB
  Correlation between right renal artery mean blood velocity (cm/sec) and CPB blood flow (L/min)
Correlation between right renal artery mean blood velocity values and CPB blood flow | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and cardiopulmonary by-pass blood flow (L/min)
Correlation between superior mesenteric artery mean blood velocity values and cardiopulmonary by-pass (CPB) blood flow | CPB 5 min: 5 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and cardiopulmonary by-pass blood flow (L/min)
Correlation between superior mesenteric artery mean blood velocity values and CPB blood flow | CPB 30 min: 30 minutes after the end of the first cardioplegia, during cardiopulmonary by-pass
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and cardiopulmonary by-pass blood flow (L/min)
Correlation between superior mesenteric artery mean blood velocity values and CPB blood flow | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and cardiopulmonary by-pass blood flow (L/min)
Correlation between right renal artery mean blood velocity values and hemodynamic parameters (mean arterial pressure, MAP) | CPB 5 min: 5 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and mean arterial pressure (mmHg)
Correlation between right renal artery mean blood velocity values and MAP | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and MAP (mmHg)
Correlation between right renal artery mean blood velocity values and MAP | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between right arterial mean blood velocity (cm/sec) and mean arterial pressure (mmHg)
Correlation between superior mesenteric artery mean blood velocity values and hemodynamic parameters (mean arterial pressure, MAP) | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and MAP (mmHg)
Correlation between superior mesenteric artery mean blood velocity values and MAP | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and mean arterial pressure (mmHg)
Correlation between superior mesenteric artery mean blood velocity values and MAP | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and MAP (mmHg)
Correlation between right renal artery mean blood velocity values and laboratory parameters (arterial PCO2) | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between right renal artery mean blood velocity (cm/sec) and arterial PCO2 (mmHg)
Correlation between right renal artery mean blood velocity values and laboratory parameters (arterial PCO2) | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and arterial PCO2 (mmHg)
Correlation between right renal artery mean blood velocity values and arterial PCO2 | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and arterial PCO2 (mmHg)
Correlation between superior mesenteric artery mean blood velocity values and laboratory parameters (arterial PCO2) | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and arterial PCO2 (mmHg)
Correlation between superior mesenteric artery mean blood velocity values and laboratory parameters (arterial PCO2) | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and arterial PCO2 (mmHg)
Correlation between superior mesenteric artery mean blood velocity values and arterial PCO2 | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and arterial PCO2 (mmHg)
Correlation between right renal artery mean mean blood velocity values and laboratory parameters (Hematocrit) | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between right renal artery mean blood velocity (cm/sec) and hematocrit
Correlation between right renal artery mean mean blood velocity values and laboratory parameters (Hematocrit) | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and hematocrit
Correlation between right renal artery mean mean blood velocity values and laboratory parameters (Hematocrit) | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and hematocrit
Correlation between superior mesenteric artery mean mean blood velocity values and laboratory parameters (Hematocrit) | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and hematocrit
Correlation between superior mesenteric artery mean mean blood velocity values and Hematocrit | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and hematocrit
Correlation between superior mesenteric artery mean mean blood velocity values and Hematocrit | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and hematocrit
Correlation between right renal artery mean blood velocity values and Temperature | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between right renal artery mean blood velocity (cm/sec) and Temperature (Celsius degrees)
Correlation between right renal artery mean blood velocity values and Temperature | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and Temperature (Celsius degrees)
Correlation between right renal artery mean blood velocity values and Temperature | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and Temperature (Celsius degrees)
Correlation between superior mesenteric artery mean blood velocity values and Temperature | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and Temperature (Celsius degrees)
Correlation between superior mesenteric artery mean blood velocity values and Temperature | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and Temperature (Celsius degrees)
Correlation between superior mesenteric artery mean blood velocity values and Temperature | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and Temperature (Celsius degrees9
Correlation between right renal artery mean blood velocity values and negative pressure applied to the venous drainage (vacuum-assist venous drainage, VAVD) | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between right renal artery mean blood velocity (cm/sec) and negative pressure applied to the venous drainage (vacuum-assist venous drainage) (mmHg)
Correlation between right renal artery mean blood velocity values and negative pressure applied to the venous drainage (vacuum-assist venous drainage, VAVD) | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and VAVD (mmHg)
Correlation between right renal artery mean blood velocity values and negative pressure applied to the venous drainage (vacuum-assist venous drainage, VAVD) | CPB 60 min: during CPB, 60 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and VAVD (mmHg)
Correlation between superior mesenteric artery mean blood velocity values and negative pressure applied to the venous drainage (vacuum-assist venous drainage, VAVD) | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between superior mesenteric artery mean blood velocity values and negative pressure applied to the venous drainage (vacuum-assist venous drainage, VAVD) (mmHg)
Correlation between superior mesenteric artery mean blood velocity values and negative pressure applied to the venous drainage (vacuum-assist venous drainage, VAVD) | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity values and negative pressure applied to the venous drainage (vacuum-assist venous drainage, VAVD) (mmHg)
Correlation between superior mesenteric artery mean blood velocity values and negative pressure applied to the venous drainage (vacuum-assist venous drainage, VAVD) | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity values and VAVD (mmHg)
Correlation between right renal artery mean blood velocity values and laboratory parameters (arterial lactate) | CPB 5 min: 5 minutes after the end of the first cardioplegia, during CPB
  Correlation between right renal artery mean blood velocity (cm/sec) and arterial lactate (mmol/L)
Correlation between right renal artery mean blood velocity values and laboratory parameters (arterial lactate) | CPB 30 min: 30 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and arterial lactate (mmol/L)
Correlation between right renal artery mean blood velocity values and laboratory parameters (arterial lactate) | CPB 60 min: 60 minutes after the end of the first cardioplegia
  Correlation between right renal artery mean blood velocity (cm/sec) and arterial lactate (mmol/L)
Correlation between superior mesenteric artery mean blood velocity and laboratory parameters (arterial lactate) | CPB 5 min: during CPB, 5 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and arterial lactate (mmol/L)
Correlation between superior mesenteric artery mean blood velocity and laboratory parameters (arterial lactate) | CPB 30 min: during CPB, 30 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and arterial lactate (mmol/L)
Correlation between superior mesenteric artery mean blood velocity and laboratory parameters (arterial lactate) | CPB 60 min: during CPB, 60 minutes after the end of the first cardioplegia
  Correlation between superior mesenteric artery mean blood velocity (cm/sec) and arterial lactate (mmol/L)
Correlation between right renal artery mean blood velocity values during CPB and Acute Kidney Injury (AKI) | CPB 5 min: during CPB, 5 minutes after the end of the first cardioplegia
  Comparison between right renal artery mean blood velocity (cm/sec) measured during CPB in patients who develop AKI according Kidney Disease Improving Global Outcomes (KDIGO) definition (AKI group) and in patients who don't develop AKI (non AKI group) during the postoperative period
Correlation between right renal artery mean blood velocity values during CPB and Acute Kidney Injury (AKI) | CPB 30 min: during CPB, 30 minutes after the end of the first cardioplegia
  Comparison between right renal artery mean blood velocity (cm/sec) measured during CPB in patients who develop AKI according KDIGO definition (AKI group) and in patients who don't develop AKI (non AKI group) during the postoperative period
Correlation between right renal artery mean blood velocity values during CPB and Acute Kidney Injury (AKI) | CPB 60 min: during CPB, 60 minutes after the end of the first cardioplegia
  Comparison between right renal artery mean blood velocity (cm/sec) measured during CPB in patients who develop AKI according KDIGO definition (AKI group) and in patients who don't develop AKI (non AKI group) during the postoperative period
Evaluation of serum Cystatin C in low right renal artery mean blood velocity during CPB | Postoperative day 1: 24 hours after the end of the cardiopulmonary by-pass
  Comparison between serum Cystatin C mean level (mg/L) measured in patients with low (below the 25th percentile) and in patients with higher (above 25th percentile) right renal artery blood velocity (cm/sec) measured during CPB
Evaluation of urinary Neutrophil Gelatinase-associated Lipocalin (uNGAL) in low right renal artery mean blood velocity | Immediate postoperative period: 4 hours after the end of the cardiopulmonary by-pass
  Comparison between urinary uNGAL mean level (ng/ml) measured immediately after surgery in patients with low (below the 25th percentile) and in patients with higher (above 25th percentile) right renal artery blood velocity (cm/sec) during CPB
Evaluation of urinary Neutrophil Gelatinase-associated Lipocalin (uNGAL) in low right renal artery mean blood velocity | Postoperative day 1: 24 hours after the end of the cardiopulmonary by-pass
  Comparison between urinary uNGAL mean level (ng/ml) measured on the first postoperative day in patients with low (below the 25th percentile) and in patients with higher (above 25th percentile) right renal artery blood velocity (cm/sec) during CPB
Evaluation of lactate in patients with low superior mesenteric artery mean blood velocity values | Immediate postoperative period: 4 hours after the end of the cardiopulmonary by-pass
  Comparison between mean arterial lactate (mmol/L) measured immediately after surgery in patients with low (below the 25th percentile) and in patients with higher (above 25th percentile) superior mesenteric artery blood velocity (cm/sec) during CPB
Evaluation of lactate in patients with low superior mesenteric artery mean blood velocity | Postoperative day 1: 24 hours after the end of the cardiopulmonary by-pass
  Comparison between arterial lactate (mmol/L) measured on the first postoperative day in patients with low (below the 25th percentile) and in patients with higher (above 25th percentile) superior mesenteric artery mean blood velocity (cm/sec) measured during CPB
Evaluation of amylase in low superior mesenteric artery mean blood velocity | Immediate postoperative period: 4 hours after the end of the cardiopulmonary by-pass
  Comparison between mean serum amylase (UI/L) measured immediately after surgery in patients with low (below the 25th percentile) and in patients with higher (above 25th percentile) superior mesenteric artery blood velocity (cm/sec) measured during CPB
Evaluation of amylase in low superior mesenteric artery mean blood velocity | Postoperative day 1: 24 hours after the end of the cardiopulmonary by-pass
  Comparison between mean serum amylase (UI/L) measured on the first postoperative day in patients with low (below the 25th percentile) and in patients with higher (above 25th percentile) superior mesenteric artery blood velocity (cm/sec) measured during CPB
Feasibility of measurement of right renal artery blood velocity during CPB | During CPB
  the number of patients in whom is possible to measure right renal artery blood velocity during CPB
Feasibility of measurement of superior mesenteric artery blood velocity during CPB | During CPB
  the number of patients in whom is possible to measure superior mesenteric artery blood velocity during CPB

CONTACTS AND LOCATIONS:
Overall Officials: Cavaliere Franco, M.D., Study Chair — Fondazione Policlinico Agostino Gemelli IRRCS
Locations (1):
- Fondazione Policlinico Universitario A,Gemelli IRCCS, Roma, Italy